CLINICAL TRIAL: NCT04496765
Title: Patients With Early-Onset Rectal Cancer Aged 40 Year or Less Have Similar Oncologic Outcomes to Older Patients Despite Presenting in More Advanced Stage; A Retrospective Cohort Study
Brief Title: Early-onset Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Other Study IDs: Mansoura2020
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- < 40 years: Patients with rectal cancer ageing 40 years or less
  Interventions: Procedure: Total mesorectal excision
- > 40 years: Patients with rectal cancer ageing more than 40 years
  Interventions: Procedure: Total mesorectal excision

INTERVENTIONS:
Procedure: Total mesorectal excision — Radical resection of rectal cancer and draining lymph nodes

SUMMARY:
The present study aimed to review the characteristics and outcome of early-onset rectal cancer in a subset of Egyptian patients aged 40 years or less. Since the previous studies assessed this point of research in CRC overall, the investigators opted to focus upon rectal cancer alone since it may represent a separate category, distinct from colon cancer, in this age group with regards to presentation, tumor behavior, and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender aged 40 years or less who presented with rectal cancer of any stage were included to the study

Exclusion Criteria:

* patients with colon cancer or other gastrointestinal cancer and patients who were lost to follow-up.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of either gender aged 40 years or less who presented with rectal cancer of any stage
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Local recurrence | 36 months after surgery
  recurrence of rectal cancer within the anatomic vicinity of the pelvis

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Study Chair — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided